CLINICAL TRIAL: NCT00029835
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multi-Center Study of Weight-Reducing Effect and Safety in Obese Patients With Untreated Dyslipidemias
Brief Title: Obese Patients With Untreated Dyslipidemias
Acronym: RIO-Lipids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4735
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Obesity; Dyslipidemia
Keywords: Obesity
MeSH Terms: conditions — Obesity; Dyslipidemias | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant (SR141716)

SUMMARY:
To assess the effect on weight loss and weight maintenance over a period of one year when prescribed with a hypocaloric diet in obese patients with untreated dyslipidemia

ELIGIBILITY:
* BMI must be greater than 27 and less than 40
* Patients with untreated dyslipidemia
* Stable weight (variation of less than 5 kg within 3 months prior to screening visit)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1033 (Actual)
Dates: Start 2001-09; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body weight at 1 year.

SECONDARY OUTCOMES:
Metabolic parameters

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (35):
- United States (28):
  - Clinic of Physicians and Surgeons, LTD, Mesa, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Irvine Center for Clinical Research (ICCR), Irvine, California
  - Los Angeles Clinical Trials, Los Angeles, California
  - Apexute, Santa Ana, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Radiant Research, Stuart, Florida
  - nTouch Research, Peoria, Illinois
  - nTouch Research, South Bend, Indiana
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Johns Hopkins Women's Research Core, Lutherville, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Twin Cities Clinical Research, Arden Hills, Minnesota
  - Radiant Research, Edina, Minnesota
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Clinical Research Services, Bismarck, North Dakota
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Division, Newtown, Pennsylvania
  - Clinical Research Center of Reading, LLC, West Reading, Pennsylvania
  - Medical University of South Carolina, Division of Clinical Pharmacology, Charleston, South Carolina
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Radiant Research, Salt Lake City, Utah
  - Clinical Research Center of Northern Virginia, Falls Church, Virginia
  - Hunter Holmes McGuire Medical Center Research Service (151), Richmond, Virginia
  - Vancouver Medical Weight Loss Clinic, Vancouver, Washington
  - Addiction & Psychiatric Medicine Research, Morgantown, West Virginia
- Sanofi-aventis Administrative Office, Macquarie Park, Australia
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Helsinki, Finland
- Sanofi-aventis Administrative Office, Milan, Italy
- Sanofi-aventis Administrative Office, Barcelona, Spain
- Sanofi-aventis Administrative Office, Bromma, Sweden
- Sanofi-aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Despres JP, Golay A, Sjostrom L; Rimonabant in Obesity-Lipids Study Group. Effects of rimonabant on metabolic risk factors in overweight patients with dyslipidemia. N Engl J Med. 2005 Nov 17;353(20):2121-34. doi: 10.1056/NEJMoa044537. PMID 16291982